CLINICAL TRIAL: NCT04686968
Title: Microfracture Combined With Suture Bridge Technique Versus Greenhouse Technique in the Treatment of Medium-sized Full-thickness Rotator Cuff Injuries: A Prospective Randomized Controlled Study
Brief Title: Microfracture Combined With Suture Bridge Technique Versus Greenhouse Technique in Treating of Rotator Cuff Injuries
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Jishuitan Hospital (Other)
Responsible Party: Principal Investigator, Chunyan Jiang, Director of Sports Medicine Service of Beijing Jishuitan hospital, Beijing Jishuitan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CJiang-Greenhouse
Record Dates: First submitted 2020-12-22; First posted 2020-12-29 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Rotator Cuff Tears; Microfractures
Keywords: rotator cuff tear; Microfractures; greenhouse; Suture Bridge Technique
MeSH Terms: conditions — Rotator Cuff Injuries; Fractures, Stress

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Greenhouse group (Experimental): Patients underwent greenhouse technique：The high-strength suture was passed through the tendon using Mason-Allen method, and then Crimson duvet procedure was performed on the foot print area from the articular surface of the humeral head to the apex of the greater tubercle. Immediately after this procedure, a lateral row anchor was used.
  Interventions: Procedure: Greenhouse Technique
- Vent group (Active Comparator): The three-line anchor suture method is the same as before, the position is between the apex of the greater tubercle and the articular surface. After the rotator cuff is sutured, the bone bed beyond the suture point to the outer edge of the greater tubercle is opened with 2.0mm Kirschner wire every 5mm ( Crimson duvet), 1cm in depth, about 6 in total.
  Interventions: Procedure: Microfracture Combined With Suture Bridge Technique

INTERVENTIONS:
Procedure: Greenhouse Technique — First, the high-strength sutures were passed through the teared tendon, and then Crimson duvet procedure was performed on the footprint from the articular margin of the humeral head to the apex of the greater tubercle, followed by a lateral row anchor.
  Arms: Greenhouse group
Procedure: Microfracture Combined With Suture Bridge Technique — A three-line anchor suture method is used as in the greenhouse technique, except that the position is between the apex of the greater tubercle and the articular surface. After the rotator cuff is sutured, the bone bed beyond the suture point to the outer edge of the greater tubercle is opened with 2.0mm Kirschner wire every 5mm ( Crimson duvet), 1cm in depth, about 6 in total.
  Arms: Vent group

SUMMARY:
Several biological augmentation procedures have recently been suggested to enhance tendon healing after Arthroscopic rotator cuff repair, such as marrow-stimulating technique with microfractures of the greater tuberosity. The purpose of this study was to introduce a new technique, "greenhouse technique", and to compare the clinical outcomes with microfracture combined with suture bridge technique.

DETAILED DESCRIPTION:
Arthroscopic rotator cuff repair has a high rate of successful subjective and functional results. Although the rate of tendon healing is reported to be around 80% for small tears, it can decrease to about 30% for large and massive tears. Poor tissue quality of bone, tendons, and muscles can affect healing and functional recovery of the rotator cuff and has been advocated as a major cause of tendon nonhealing and/or retear. Several biological augmentation procedures have recently been suggested to enhance tendon healing after Arthroscopic rotator cuff repair, such as marrow-stimulating technique with microfractures of the greater tuberosity. The purpose of this study was to introduce a new technique, "greenhouse technique", and to compare the clinical outcomes with microfracture combined with suture bridge technique.

ELIGIBILITY:
Inclusion Criteria:

* Medium-sized full-thickness rotator cuff tear confirmed during shoulder arthroscopy
* Between 20-65 years old

Exclusion Criteria:

* Bilateral rotator cuff tear
* Underwent ipsilateral surgery
* Large-to-massive rotator cuff tear
* Combined with Bankart, SLAP or AC lesion
* Combined with diabetes, smoking, immune disease, osteoporosis, and large nodular cystic degeneration

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2021-07 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
American Shoulder and Elbow Surgeons Shoulder (ASES) score | 1 year postoperatively
  A patient-reported outcome uesed to assess the shoulder function,range 0-100, higher scores mean a better outcome
American Shoulder and Elbow Surgeons Shoulder (ASES) score | 2 years postoperatively
  A patient-reported outcome uesed to assess the shoulder function,range 0-100, higher scores mean a better outcome
tendon integrity | 1 year postoperatively
  MRI was used to assess the integrity of the repaired rotator cuff tendon
Visual Analogue Scale(VAS) | 1 year postoperatively
  A patient-reported outcome uesed to assess pain severityrange 0-10, higher scores mean a worse outcome
Visual Analogue Scale(VAS) | 2 year postoperatively
  A patient-reported outcome uesed to assess pain severityrange 0-10, higher scores mean a worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Chunyan Jiang, M.D., Principal Investigator — Sports Medicine Service, Beijing Jishuitan hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Milano G, Saccomanno MF, Careri S, Taccardo G, De Vitis R, Fabbriciani C. Efficacy of marrow-stimulating technique in arthroscopic rotator cuff repair: a prospective randomized study. Arthroscopy. 2013 May;29(5):802-10. doi: 10.1016/j.arthro.2013.01.019. Epub 2013 Mar 21. PMID 23522987
- [Background] Kim C, Lee YJ, Kim SJ, Yoon TH, Chun YM. Bone Marrow Stimulation in Arthroscopic Repair for Large to Massive Rotator Cuff Tears With Incomplete Footprint Coverage. Am J Sports Med. 2020 Nov;48(13):3322-3327. doi: 10.1177/0363546520959314. Epub 2020 Sep 25. PMID 32976717
- [Background] Taniguchi N, Suenaga N, Oizumi N, Miyoshi N, Yamaguchi H, Inoue K, Chosa E. Bone marrow stimulation at the footprint of arthroscopic surface-holding repair advances cuff repair integrity. J Shoulder Elbow Surg. 2015 Jun;24(6):860-6. doi: 10.1016/j.jse.2014.09.031. Epub 2014 Dec 2. PMID 25487905